CLINICAL TRIAL: NCT04626388
Title: Postoperative Score Predictive of the Prognosis of Acetabular Fractures
Acronym: SCORE_COTYLE
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: SCORE_COTYLE
Record Dates: First submitted 2020-11-10; First posted 2020-11-12 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-04

CONDITIONS: Acetabular Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acetal fractures are joint fractures that occur in the hip. These fractures affect the functional prognosis of the hip in the short, medium and long term. In the acetabulum fractures operated on, there is a radiological score in the literature allowing the prognosis to be predicted depending on the quality of the postoperative reduction. This score is based on the quality of postoperative reduction assessed on pelvic radios. In addition, the thresholds for poor / good results were determined empirically.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient operated on for an acetabular fracture at the GHPSJ between January 2004 and December 2014
* Patient with a minimum postoperative follow-up of 2 years
* French-speaking patient

Exclusion Criteria:

* Patient treated conservatively.
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection
* Patient objecting to the use of his medical data as part of this study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients were operated on for an acetabulum fracture within the Paris Saint Joseph Hospital Group, between January 2004 and December 2014, with a minimum post-operative follow-up of 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Total hip replacement | Year 2
  This ouctome corresponds to the total hip prosthesis.

SECONDARY OUTCOMES:
Post-operative complications | Year 2
  This ouctome corresponds to the postoperative complication rate.
Delay of total hip replacement | Year 2
  This ouctome corresponds to the delay of total hip replacement.

CONTACTS AND LOCATIONS:
Overall Officials: Elias MELHEM, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Result] Matta JM, Mehne DK, Roffi R. Fractures of the acetabulum. Early results of a prospective study. Clin Orthop Relat Res. 1986 Apr;(205):241-50. PMID 3698383
- [Result] Matta JM. Fractures of the acetabulum: accuracy of reduction and clinical results in patients managed operatively within three weeks after the injury. J Bone Joint Surg Am. 1996 Nov;78(11):1632-45. PMID 8934477
- [Result] Verbeek DO, van der List JP, Villa JC, Wellman DS, Helfet DL. Postoperative CT Is Superior for Acetabular Fracture Reduction Assessment and Reliably Predicts Hip Survivorship. J Bone Joint Surg Am. 2017 Oct 18;99(20):1745-1752. doi: 10.2106/JBJS.16.01446. PMID 29040129
- [Result] Jouffroy P, Sebaaly A, Aubert T, Riouallon G. Improved acetabular fracture diagnosis after training in a CT-based method. Orthop Traumatol Surg Res. 2017 May;103(3):325-329. doi: 10.1016/j.otsr.2016.10.020. Epub 2016 Dec 23. PMID 28017876
- [Result] Verbeek DO, van der List JP, Moloney GB, Wellman DS, Helfet DL. Assessing Postoperative Reduction After Acetabular Fracture Surgery: A Standardized Digital Computed Tomography-Based Method. J Orthop Trauma. 2018 Jul;32(7):e284-e288. doi: 10.1097/BOT.0000000000001161. PMID 29481491